CLINICAL TRIAL: NCT00256529
Title: Prospective Analysis of Eosinophilic Esophagitis in Patients Presenting With Dysphagia
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Kathryn A. Peterson, MD, University of Utah
Other Study IDs: 14543
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2014-12-15 (Estimated); Status verified 2014-12

CONDITIONS: Esophagitis
Keywords: dysphagia; eosinophilic esophagitis
MeSH Terms: conditions — Esophagitis; Deglutition Disorders; Eosinophilic Esophagitis | interventions — Endoscopy, Digestive System; Biopsy; Gastroscopy

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 4 quadrant distal and proximal biopsies of the esophagus
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- I: All subjects presenting in with dysphagia will be in this cohort.
  Interventions: Procedure: EGD with biopsies

INTERVENTIONS:
Procedure: EGD with biopsies — All subjects presenting with dysphagia will undergo an EGD with distal and proximal biopsies of the esophagus.
  Other Names: Upper endoscopy

SUMMARY:
This is a prospective descriptive cross sectional study to determine the percentage of patients presenting with dysphagia who are found to have eosinophilic esophagitis (EoE) and to establish which presenting factors warrant esophageal biopsies. We hypothesize that a greater than expected percentage of patients who are biopsies will have histologic changes consistent with EE.

DETAILED DESCRIPTION:
All patients presenting with dysphagia who do not already carry a previous diagnosis for their dysphagia will be asked to enroll. If patients have undergone previous work up for dysphagia such as manometry, 24-hour probe, or barium swallow they can still participate in this study. Informed consent will take place prior to enrollment. After patients present with dysphagia they will fill-out a questionnaire regarding their dysphagia symptoms. An EGD with biopsies will then be performed. Biopsies will be taken from 4 quadrants in the proximal and distal esophagus. The distal esophagus biopsies will be taken 5 cm proximal to the Z-line. Proximal biopsies will be taken anywhere proximal to 30 cm from the incisors.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-90 presenting with dysphagia or food impaction
* Ability to undergo esophagogastroduodenoscopy and biopsies
* No significant cardiopulmonary disease, or other contraindication to EGD

Exclusion Criteria:

* Contradiction to EGD and/or biopsies such as Boerhaave's syndrome, or history or bleeding disorder or elevated INR
* Inability to provide informed consent
* Esophageal varices

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting with dysphagia will be eligibile for enrollment into the study.
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2005-11; Primary Completion 2011-07 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To assess the percentage of patients who present with dysphagia who have EE by histologic criteria | December 2010

SECONDARY OUTCOMES:
To assess the demographics of the EE patients with dysphagia | December 2010
To measure the frequency, severity, and time course of dysphagia in patients with EE | December 2010
To assess percentage of EE patients with recurrent, versus acute dysphagia | December 2010

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Byrne, M.D., Principal Investigator — University of Utah
Locations (1):
- Department of Veterans Affairs, Salt Lake City, Utah, United States